CLINICAL TRIAL: NCT05898633
Title: Phase 1 Safety Trial of Recombinant Surfactant Protein D to Prevent Neonatal Chronic Lung Disease
Brief Title: Recombinant Surfactant Protein D (rfhSP-D) to Prevent Neonatal Chronic Lung Disease
Acronym: RESPONSE
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: Medical Research Council (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18/0564; 2021-001824-16 (EudraCT Number)
Record Dates: First submitted 2023-03-24; First posted 2023-06-12 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Chronic Lung Disease of Prematurity; Respiratory Distress Syndrome in Premature Infant; Bronchopulmonary Dysplasia
Keywords: Preterm Infants; Recombinant Surfactant Protein D
MeSH Terms: conditions — Bronchopulmonary Dysplasia

STUDY DESIGN:
Intervention Model Description: A Bayesian Continual Reassessment Method (CRM) will be used for the RESPONSE trial to inform how the IMP dose should be adapted for the next cohort based on past trial data. The CRM is a model-based design that uses a statistical model to estimate the risk of dose limiting events (DLE) per dose level. The target level of DLEs is set at 20% The CRM model does not allow dose-skipping. The recommended phase 2 dose in terms of safety (efficacy will also be taken into account) will be the highest dose level that has an estimated probability of DLE closest but below the target DLE level of 20%.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Recombinant fragment of human surfactant protein D (rfhSP-D) administration (Experimental): This is a single arm trial with administration of rfhSP-D.
  All participants will be administered rfhSP-D via an endotracheal tube in 1-3 doses in the first 24-48hrs after birth whilst the infant is still intubated and ventilated.
  A dose escalation design from 1mg/kg to 4mg/kg will be used. Infants are enrolled in cohorts of three, with the first cohort receiving the lowest dose 1mg/kg.
  Participants are followed up until they are discharged from hospital.
  Interventions: Drug: Recombinant fragment of human surfactant protein D (rfhSP-D)

INTERVENTIONS:
Drug: Recombinant fragment of human surfactant protein D (rfhSP-D) — Administration of rfhSP-D
  Other Names: rfhSP-D

SUMMARY:
The purpose of this study is to identify the safest dose of recombinant surfactant protein D (drug name: rfhSP-D) that can be administered to preterm infants born at less than 30 weeks gestation, and to help identify whether this can prevent the development of neonatal chronic lung disease.

DETAILED DESCRIPTION:
This is a Phase I, dose escalation safety study that aims to identify the recommended phase 2 dose of recombinant fragment of human surfactant protein D (rfhSP-D) (drug name: rfhSP-D) for infants at risk of neonatal chronic lung disease. This study will aim to establish if the administration of rfhSP-D to the lungs of preterm babies, via an endotracheal tube, is safe at the proposed dosage range (1mg/kg - 4mg/kg) and whether this dose results in detectable concentrations in lung secretions or serum.

Surfactant protein D (SP-D) is a naturally occurring component of the surfactant system with anti-inflammatory properties. Current surfactant replacement therapy contains phospholipids and surfactant proteins B and C (SP-B and SP-C) but no surfactant protein A (SP-A) or surfactant protein D (SP-D).

Proof of concept regarding the anti-infective and anti-inflammatory activity of SP-D has been achieved in mouse and a preterm lamb models of lung disease and supports increasing evidence of the role played by deficiency of SP-D in human respiratory diseases.

Subjects will be enrolled in cohorts with increasing dose. Whether or not the dose is escalated will depend on the occurrence of dose limiting events (DLE) in all current patients and the doses that they have received. A model will be used to estimate the risk of DLE per dose level. Initial estimates of these risks will be updated using data collected throughout the trial.

Up to 24 infants of less than 30 weeks gestation will be recruited in the study and receive intra-tracheal administration of SP-D59, in the dose range 1mg/kg, 2mg/kg or 4mg/kg per dose for up to 3 doses. The first dose of SP-D59 will be given as soon as possible after the first dose of standard surfactant therapy (e.g., Curosurf). Subsequent doses of the IMP will be given at 12 hours and 24 hours after the first dose was administered.

ELIGIBILITY:
Participant Inclusion Criteria:

1. Inborn infants born at between 23 weeks and 0 days and 29 weeks and 6 days gestation.
2. Infant must be intubated or planned to be intubated for respiratory distress at time of eligibility check, and this should be done within 12 hours from time of birth.
3. Receiving standard surfactant therapy
4. Clinically stable on mechanical ventilation. Stability is defined at the time of IMP instillation and is defined below.
5. Written informed consent from parents/guardians/person with legal responsibility

Definition of stability:

1. Blood gases within the normal range for preterm infants (pH>7.20; paCO2 <60mmHg)
2. Mean blood pressure with or without inotropic support at at least gestational age or above (mmHg)
3. No evidence of a pneumothorax
4. Clinical observations within acceptable range for an infant of that gestational age
5. No stability concerns from the attending neonatologist

Participant Exclusion Criteria:

1. Congenital anomalies i.e any major antenatal diagnosed congenital abnormalities such as congenital heart disease, suspected or known chromosomal abnormalities
2. Parents/legal guardians unable to give consent due to learning or other difficulties
3. Infants requiring only CPAP support without the need for surfactant replacement therapy, i.e. without endotracheal intubation
4. Infants born in very poor condition and judged too sick or unstable to be included (high risk of mortality) in an experimental first in human study, for example infants that are requiring maximal intensive care therapy and have findings such as a grade IV intraventricular haemorrhage that is likely to be life limiting.
5. Infants that are born out of the participating site.
6. Participation in any other interventional study (participation in an observational study is permissible).

Ages: 23 Weeks to 30 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Estimated)
Dates: Start 2024-04-06 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Occurence of Dose Limiting Events to assess the safety profile of the IMP (rfhSP-D) | Day 0 to 96 hours
  To assess the safety profile of rfhSP-D across dose levels based on the occurrence of Dose Limiting Events (DLEs) which are events Garde 3 or above on the NAESS scale related to the IMP
To find recommended Phase 2 Dose of rfhSP-D | Day 0 to the point of hospital discharge (40 weeks post-menstrual age)
  To establish the Recommended Phase 2 Dose (RP2D) of rfhSP-D for preterm infants born at gestational age of 23 weeks to 29 weeks + 6 days.

SECONDARY OUTCOMES:
Occurrence of non-dose limiting events, including SAE/AEs | Day 0 to the point of hospital discharge (40 weeks post-menstrual age)
  To establish the safety profile of rfhSP-D across dose levels based on the occurrence of non-DLEs, including SAE/AEs.
Systemic absorption of rfhSP-D | Day 0 to 36 weeks post menstrual age
  To evaluate systemic absorption of rfhSP-D using serial measurements of rfhSP-D in serum and its continued presence in tracheal fluid.
Effects of rfhSP-D on the cell counts of inflammatory markers | Day 0 to 36 weeks post menstrual age
  To determine the effect of rfhSP-D on Inflammatory markers in the lung secretions (eg.cell counts of the following markers: neutrophils, macrophages, MMPs, neutrophil elastase, IL-8,IL-6, IL-1).

CONTACTS AND LOCATIONS:
Overall Officials: Howard Clark, MBBS, Principal Investigator — University College London Hospital
Locations (1):
- University College London Hospitals, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
There is currently no plan to make individual participant data available to other researchers. Written requests will be considered by the RESPONSE Trial Management Group.

REFERENCES:
- [Derived] Bhatt R, Madsen J, Castillo-Hernandez T, Chant K, Dehbi HM, Marlow N, Clark H. Recombinant fragment of human surfactant protein D to prevent neonatal chronic lung disease (RESPONSE): a protocol for a phase I safety trial in a tertiary neonatal unit. BMJ Open. 2024 Aug 17;14(8):e086394. doi: 10.1136/bmjopen-2024-086394. PMID 39153779